CLINICAL TRIAL: NCT00082095
Title: A Randomized, Open-Label Trial Comparing Treatment With Either Pegylated Liposomal Doxorubicin or Capecitabine as First Line Chemotherapy for Metastatic Breast Cancer in Women 60 Years and Older
Brief Title: To Compare Treatment With Doxorubicin or Capecitabine for Metastatic Breast Cancer in Women 60 Years and Older
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to poor recruitment (after enrolling 62 of planned 300 patients in 20 months
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004645; DO03-21-022 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2004-04-29; First posted 2004-04-30 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Breast Cancer; Pegylated Liposomal Doxorubicin; Capecitabine; DOXIL; Xeloda
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (doxorubicin) (Experimental): Pegylated liposomal doxorubicin 40 mg/m2 administered intravenously on Day 1 of each cycle. Cycle is repeated every 28 days, up to one year.
  Interventions: Drug: Pegylated liposomal doxorubicin
- Group 2 (capecitabine ) (Active Comparator): Capecitabine administered orally at a dosage of 2000 mg/m2/day (1000 mg/m2 BID) for 14 consecutive days followed by a 7-day rest period. Cycle is repeated every 21 days, up to one year.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — Type=exact number, unit=mg/m2, number=40, form=infusion, route=intravenous. Pegylated liposomal doxorubicin will be administered on Day 1 of each cycle. Cycle will be repeated every 28 days, up to 1 year.
  Other Names: DOXIL
  Arms: Group 1 (doxorubicin)
Drug: Capecitabine — Type=exact number, unit=mg, number=500, form=tablet, route=oral. Capecitabine will be administered at a dosage of 1000 mg/m2 twice daily for 14 consecutive days followed by a 7-day rest period. Cycle is repeated every 21 days, up to one year.
  Other Names: Xeloda
  Arms: Group 2 (capecitabine )

SUMMARY:
The main purpose of this study is to compare treatment with either pegylated liposomal doxorubicin or capecitabine as first line chemotherapy for metastatic breast cancer in women 60 years and older.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), multicenter study comparing with pegylated liposomal doxorubicin (PLD) with capecitabine as first line chemotherapy of metastatic breast cancer in women 60 years and older. The study consists of a screening Phase (up to 14 days prior to treatment), treatment phase (up to 1 year), and post-treatment follow-up phase. The planned duration of treatment was 1 year in the absence of disease progression or unacceptable toxicity. Approximately 300 patients will be enrolled and randomly assigned to receive 1 of 2 treatment groups (PLD or capecitabine). Safety evaluations will consist of vital sign examination, physical examination, incidence and severity of adverse events, and laboratory tests findings and will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or pathologically proven metastatic breast cancer
* Eastern Cooperative Oncology Group performance status between 0-2
* Adequate bone marrow, renal and liver functions within normal limits
* Left ventricular ejection fractions more than 45% measured by multiple gated acquisition scan or echocardiogram within 6 weeks of randomization

Exclusion Criteria:

* Prior chemotherapy for metastatic disease (hormonal or chemotherapy in adjuvant setting and hormonal therapy in metastatic setting is allowed)
* Prior treatment with capecitabine or pegylated liposomal doxorubicin in the adjuvant setting (prior anthracyclines up to certain dose limit is allowed)
* Evidence of brain metastases unless previously treated and asymptomatic for 3 months or greater
* History of cardiac disease with New York Heart Association Class II or greater or clinical evidence of congestive heart failure
* Anthracycline resistant disease (locally recurrent or metastatic disease while on adjuvant anthracycline therapy or relapse less than 18 months after therapy completion)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Time to disease progression | Up to disease progression or death
  Time to disease progression is the duration in months from the date of randomization to the first documented evidence of disease progression or death caused by disease progression before the end of study. Time to disease progression will be compared between patients treated with doxorubicin and capecitabine.

SECONDARY OUTCOMES:
Overall Response rate | Up to disease progression or death
  Overall response rate is measured as the number of patient with complete and partial responses. It will be compared between patients treated with doxorubicin and capecitabine.
Overall survival | Up to 2 years after last patient is enrolled or death
  Overall survival is the duration from date of randomization to the date of death due to any cause during the study. It will be compared between patients treated with doxorubicin and capecitabine.
Number of patients with adverse events | Up to 1 month after intake of last dose of study medication
  Safety evaluated as "number of patients with adverse events" is compared between 2 treatment groups (doxorubicin and capecitabine).
The European Organization for Research and Treatment of Cancer (EORTC) QLQ (Quality of Life Questionnaire) - C30 | Day 1 and end of treatment
  The 30 item questionnaire to assess quality of life incorporates five functional scales: general physical symptoms, physical functioning, psychological distress, social functioning, and fatigue/malaise. Most items are rated on a 4 point Likert scale ranging from 0 = "not at all" to 4 = "very much". The effect of doxorubicin and capecitabine on the quality of life measured by the EORTC QLQ-C30 is assessed.
Subjective Significance Questionnaire (SSQ) | Day 1 and end of treatment
  The SSQ consists of 4 items in which patients rate the degree to which they experienced an improvement or deterioration in their physical condition, emotional state, ability to enjoy their social life, and overall quality of life since there last QOL assessment.Each of the four items are rated on a 7 point Likert scale ranging from 0 = "very much worse" to 7 = "very much better". The effect of doxorubicin and capecitabine on the quality of life measured by the SSQ is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (27):
- United States (27):
  - Fountain Valley, California
  - Oxnard, California
  - Soquel, California
  - Boca Raton, Florida
  - New Port Richey, Florida
  - Plantation, Florida
  - Atlanta, Georgia
  - Springfield, Illinois
  - Hazard, Kentucky
  - Shreveport, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Clinton Township, Michigan
  - Saint Louis Park, Minnesota
  - Lebanon, New Hampshire
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - Armonk, New York
  - New City, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Fort Worth, Texas
  - Fredericksburg, Texas
  - Burlington, Vermont
  - Colchester, Vermont
  - Everett, Washington
  - Vancouver, Washington

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- See also: A Randomized, Open-Label Trial Comparing Treatment with Either Pegylated Liposomal Doxorubicin or Capecitabine as First Line Chemotherapy for Metastatic Breast Cancer in Women 60 Years and Older — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=613&filename=CR004645_CSR.pdf